CLINICAL TRIAL: NCT05142254
Title: A Randomized Controlled Double-Blind Trial for Prevention of Recurrent Ischemic Priapism in Men With Sickle Cell Disease: A Pilot Study
Brief Title: A Trial for Prevention of Recurrent Ischemic Priapism in Men With Sickle Cell Disease: A Pilot Study
Acronym: PIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael DeBaun, M.D. MPH, Director Vanderbilt-Meharry Center for Excellence in Sickle Cell Disease, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202504
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Priapism Due to Sickle Cell Disease
MeSH Terms: interventions — Tadalafil; Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Double-Blind Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The primary study statistician will be supported by a local statistician in Nigeria to perform the randomization process. After the random allocation, all study personnel and participants will be blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tadalafil and Hydroxyurea (Experimental): Tadalafil 2.5-5 mg/day and Hydroxyurea 20 mg/kg/day
  Interventions: Drug: Tadalafil; Drug: Hydroxyurea
- Placebo and Hydroxyurea (Placebo Comparator): Placebo and Hydroxyurea 20 mg/kg/day
  Interventions: Drug: Hydroxyurea; Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — 2.5-5 mg/day
  Arms: Tadalafil and Hydroxyurea
Drug: Hydroxyurea — 20 mg/kg/day
Drug: Placebo — identical placebo to tadalafil created by Bond Biochemical, who is manufacturing the tadalafil as well.
  Arms: Placebo and Hydroxyurea

SUMMARY:
To conduct a randomized controlled internal pilot feasibility trial for the prevention of recurrent ischemic priapism referred to as the Priapism in Nigeria (PIN) trial. The study team will enroll a minimum of 30 participants and a maximum of 200 participants. Study investigators hypothesize that hydroxyurea therapy combined with tadalafil is superior to a combination of hydroxyurea and placebo in the prevention of recurrent ischemic priapism.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is one of the commonest genetic diseases in the world. Approximately 300,000 newborns are born with SCD every year, with 50% of the birth being in Nigeria alone. This huge burden makes Nigeria critical to any intervention that seeks to address the challenges of individuals with SCD. Men with SCD experience many complications, which can even affect their sexuality and reproductive health. One of the most common, but often neglected complications of SCD in men is priapism. Priapism is defined as a painful, purposeless, and sustained erection. In men with SCD, priapism tends to be recurrent and devastating. The prevalence of priapism was 42% in Jamaican men with SCD. Researchers reported the incidence of priapism in SCD to be very low before the age of 10 years, but the cumulative incidence rose to 32.7% by the age of 20 years. Researchers reported the prevalence of priapism in SCD to be 35%, out of which 72% was recurrent ischemic priapism (lasting <4 hours). The majority of the individuals with SCD experienced their first episode of priapism before the age of 20 years, with a mean age of onset being 15 years. In a cross-sectional study of 353 men with SCD, conducted by our team in Kano, Nigeria, the prevalence of priapism was approximately 32%; out of which 74% was recurrent ischemic priapism. In the same study, the prevalence of priapism in men without SCD (n=250) was 2%. The results from focus groups (3 in Nigeria and 3 in the U.S.) our team conducted revealed men with SCD who experienced recurrent ischemic priapism struggled with embarrassment, shame, anxiety and depression, and declining sexual function.

The prevention and treatment of ischemic priapism in SCD is still inadequate. Researchers used a combination of preventive oral etilefrine and self-administered intracavernosal injection of etilefrine for breakthrough priapism lasting >1 hour. Sixty-six percent (4 of 6) had no recurrence of priapism while the remaining two used intracavernosal injection of etilefrine. In a non-RCT study, Researchers reported a good response to oral etilefrine; which was shown to have reduced the frequency of recurrent ischemic priapism in SCD (mean difference 5.78); P < 0.0001.(21) However, in the only RCT for this drug, etilefrine was found to have no efficacy over placebo. Researchers showed that in 35 patients on graded doses of finasteride (5-alpha reductase inhibitor), priapism recurrences were reduced from an average of 22.7 to 2.1 at the end of the 120-day follow-up. A combination of oral ketoconazole with prednisolone showed a promising result in case-series reported by researchers. However, an RCT (n=40) showed no efficacy of ketoconazole (81.25% and 83% in both arms still having post-operative painful erections). In another study, hydroxyurea was shown to have decreased priapism recurrences in 4 of 5 men treated with a high dose. Nonetheless, stopping hydroxyurea heralded relapse of priapism. Researchers reported that sildenafil has controlled priapism experiences in 6 of 7 men observed. Non-RCT designs, small sample sizes, or adverse effects of the trial medications limit most of these studies.

This conceptual framework is based on the synergistic effect of tadalafil (PDE-5 inhibitor, which increases the bioavailability of cGMP), and hydroxyurea (NO donor). In SCD there is chronic hemolysis causing depletion of NO and dysregulation of PDE-5, which underpin the molecular basis of priapism. Chronic dosing of low-dose tadalafil inhibits PDE-5 to paradoxically restore the normal homeostatic mechanism of the NO-cGMP-PDE-5 pathway. Restored PDE-5 function helps prevent recurrent ischemic priapism. Despite the need, all prior priapism studies did not provide sufficient evidence for practice-based outcomes. Several reasons exist for the lack of any substantial progress for secondary prevention of ischemic priapism, the foremost of which is that SCD is a rare disease in high-income settings where most of the studies have been conducted. To overcome these limitations, the investigators propose an internal pilot trial to assess the feasibility trial in a setting where there are over 5000 men available to be enrolled in one city, Kano Nigeria. The trial will also build on the infrastructures and workflow established by NIH-funded pre-existing SCD stroke prevention trials conducted at the same hospitals in Kano.

The aims are:

1. To conduct a randomized controlled internal pilot trial for prevention of recurrent ischemic priapism (hydroxyurea + tadalafil vs hydroxyurea + placebo), referred to as the Priapism in Nigeria (PIN) trial.

   Outcomes: The focus of this internal pilot feasibility trial is not to determine efficacy. Rather the focus is on the recruitment, retention, and adherence rate of therapy. However, we intend to have preliminary findings that will guide us about the likelihood of efficacy of the intervention. Thus, our secondary clinical outcome will be a reduction in the recurrence rate of priapism. Our secondary outcome will be the improvement of erectile and sexual functions based on high scores on IIEF and PROMIS questionnaires. Sample Size: 100
2. To assess the effect of moderate-dose hydroxyurea on spermatogenesis.

   Outcomes: Prior clinical trials have shown hydroxyurea to be safe even in sub-Saharan Africa where the rate of infections is high; however, there is a growing concern for its relative safety in men based on its potentially damaging effect on spermatozoa. Therefore, all participants will have seminal fluid collected and assessed at baseline according to the World Health Organization (WHO) standard using the SQA IIC-P auto-analyzer. Repeat semen assessments will be done at intervals of 12 months (completion of the trial), and at 3 months post completion of the trial. Semen Collection: The participants will be given a paper containing clear step-by-step instructions for semen collection, including abstinence from sex and masturbation for 4 days before the collection date. No use of condom, oral, or vaginal sex for semen collection to avoid contamination. Semen collection will be by masturbation. To ease masturbation, a penile vibrating stimulation (PVS) device will be provided at the collection point. Sample size: The same number of participants (n=100) included in the Aim 1 above (internal pilot feasibility trial)
3. To follow up participants with priapism, who are ineligible for inclusion in the feasibility trial, under the standard of care cohort. Outcomes: We will assess for all outcomes as in Aim1. Sample size: we estimate that about 50% of the participants who consented for the study may be ineligible for some of the stated criteria. Thus, we plan to include about 50 participants in this cohort.

Sample size determination: For the internal pilot feasibility trial (Aim 1), our main focus is whether or not this trial is feasible based on recruitment, retention, and adherence rates to trial therapy. We will assume a binomial distribution and calculate the corresponding one-sided 95% confidence intervals. With a sample size of 100, using the Clopper-Pearson formula, with expected retention rates of 80% in each group, and with observed compliance rates of 87% and higher, we obtain a lower bound on compliance of 75.0%.

Analysis plan: For aim 1, we will use proportions and confidence intervals to calculate the percentages of participants who have agreed to participate in the trial, adhere to trial drugs and stay to complete the one-year follow-up. We will use negative binomial regression to calculate the hazard rate for rate of priapism recurrence in both arms and determine whether there is a difference in recurrence between the two arms. We will use multiple imputation analyses for missing data. Adverse side effects will be reported as proportions with 95% confidence intervals and compared between the two groups using the Chi-Square test. In contrast, rates of penile aspirations will be compared using negative binomial regression. We will also use a non-parametric test (Mann Whitney U) and negative binomial regression to compare hospitalizations for acute pain between the 2 arms of the trial, controlling for age and other baseline characteristics. For aim 2, we will use paired t-test or non-parametric equivalent to calculate the mean difference in total sperm counts at discrete time points. For aim 3, we will not do power analysis since this is an exploratory study.

During study visits, we will also systematically collect data on potential side effects of tadalafil using National Cancer Institutes (NCI) Patient-Reported Outcomes- Common Terminology Criteria for Adverse Events (PRO-CTCAE). Data on serious adverse effects such as mortality will also be collected and analyzed. Data on participants developing major priapism necessitating surgical interventions (penile aspirations and shunt surgery) will be collected for comparison between two arms of the trial. All data on tadalafil's adverse effects will be reviewed weekly to provide a guide on whether the trial should progress or be halted by the Principal Investigator or Data Safety Monitoring Board (DSMB).

Our strategy to ensure the retention of participants in the trial will include collecting the phone numbers of each participant and at least two people who are very close to the participant (whom we can call whenever we cannot find the participant). We will make phone calls every week to remind the participants about adherence to the therapies and study visits. Compensation will be given to participants for their study visits. These data will be collected locally, and not included at the Data Coordinating Center (VUMC). Outcomes: The focus of this internal pilot feasibility trial is not to determine efficacy. Rather the focus is on the recruitment, retention and adherence rate of therapy. However, we intend to have preliminary findings that will guide us about the likelihood of efficacy of the intervention. Thus, our secondary clinical outcome will be a reduction in the recurrence rate of priapism. Our secondary outcome will be the improvement of erectile and sexual functions based on high scores on IIEF and PROMIS questionnaires.

Trained study personnel will approach the eligible participants for consenting. After obtaining signed informed consent and ensuring they have fulfilled inclusion criteria, the participants will be randomized 1:1 to the treatment and placebo arms. The primary study statistician will be supported by a local statistician in Nigeria to perform the randomization process. After the random allocation, all study personnel and participants will be blinded to the treatment. The treatment arm will include tadalafil, given orally initially at a low-dose of 2.5 mg daily for four weeks. If tolerated very well during the four weeks, the dose will be increased to 5.0 mg daily as the final dose. Tadalafil and the identical placebo will be purchased from a local pharmaceutical company, Bond Chemical Nigerian Limited, which is licensed to produce tadalafil and hydroxyurea in Nigeria. Participants will be instructed to take tadalafil or placebo in the morning for this trial. Chronic morning dosing with tadalafil will allow the drug to be metabolized and is unlikely to be associated with sleep-related erections. Both treatment and placebo arms will be on hydroxyurea as standard care. Hydroxyurea will be given orally at a moderate-dose of 20mg/kg/day and is also produced by the Bond Chemical Nigerian Limited. The moderate-dose of hydroxyurea is found to be effective, with minimal adverse effects, in the preliminary data of stroke prevention in Nigeria (1R01NS094041) trial just recently completed in Kano, Nigeria. Both arms of the trial will be followed for one year; afterward, the trial will go into the open-label phase. The participant can select whether they want to continue either therapy or start a new treatment. At the baseline, demographic and clinical data from medical records of the participants will be collected. The data will include but are not limited to: co-morbidities (hypertension, diabetes, etc.), drug history (antihypertensives, aphrodisiacs, hormonal shots, alpha receptor agonists, antipsychotics, etc.), pain history, and blood transfusions history. The investigators will use internationally validated questionnaires (International Index of Erectile Function [IIEF], PROMIS Erectile function, sexual activity, and satisfaction with sex life) to evaluate erectile and sexual functions of the participants at baseline and subsequent follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Men with confirmed diagnosis of HbSS or Hb beta zero thalassemia
* Ages between 18 to 40 years
* Eligible study participants must receive care in an SCD clinic at AKTH and MMSH at the time of the recruitment
* Participants must commit to long-term follow-up and taking the trial medications
* At least 3 episodes of priapism, each lasting for no less than an hour in the past 6 months.
* Adequate renal and hepatic function (baseline liver enzymes and synthetic activities should be no more than four-fold above the reference ranges for Aminu Kano Teaching Hospital (AKTH). These are the ranges obtained in AKTH: Alkaline phosphatase: 42-110 U/L, Alanine transaminase: 4-34 U/L, Aspartate transaminase: 7-45 U/L, Albumin: 32-52 g/L, and Globulin: 32-43 g/L.

Exclusion Criteria:

* Individuals already enrolled in another clinical trial
* eGFR <50ml/min
* Liver cirrhosis based on clinical history, laboratory data or both
* Previously known pulmonary hypertension based on TRJV greater than 3.0 m/sec
* Contraindications to tadalafil (arrhythmia, severe liver disease, concurrent use of nitrates, etc.) or hydroxyurea (leg ulcer, hypersensitivity, etc.).
* Patients who have penile prosthetic implants or shunts or any other surgical procedure on the penis
* Patients who have taken drugs/medications that may induce priapism over the 14 weeks before trial:
* Medications injected directly into the penis to treat erectile dysfunction, such as alprostadil, papaverine, phentolamine, and others
* Antidepressants, such as fluoxetine, bupropion, and sertraline
* Alpha blockers including prazosin, terazosin, doxazosin, and tamsulosin
* Medications used to treat anxiety or psychotic disorders, such as hydroxyzine, risperidone, olanzapine, lithium, clozapine, chlorpromazine, and thioridazine
* Blood thinners, such as warfarin and heparin
* Hormones such as testosterone or gonadotropin-releasing hormone
* Medications used to treat attention-deficit/hyperactivity disorder (ADHD), such as atomoxetine (Strattera)
* Alcohol, marijuana, cocaine and other illicit drug abuse can cause priapism
* Not able to understand or comply with study instructions and requirements

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
A change in the recurrence rate of priapism | Within a year, we will measure recurrence rates
  We will use negative binomial regression to calculate the hazard rate for rate of priapism recurrence in both arms and determine whether there is a difference in recurrence between the two arms.

SECONDARY OUTCOMES:
The rate of vaso-occlusive pain, including hospitalizations | Baseline- one year
  We will use a non-parametric test (Mann Whitney U) and negative binomial regression to compare hospitalizations for acute pain between the 2 arms of the trial, controlling for age and other baseline characteristics.
Change of erectile and sexual functions | Baseline- one year
  International Index of Erectile Function (IIEF) Survey- 15 questions on a scale from 0 to 5. The survey examines 4 main domains of male sexual function and overall satisfaction. The maximum total score for the survey is 75, with each domain having a maximum score of 30, 10, 10, 15, and 10 respectively . Scores below 14 in the first domain (out of 30) indicate erectile function issues.
Change of erectile and sexual functions | Baseline- one year
  Promis Bank V20 Satisfaction With Sex Life (5 total questions, ranging from not at all to very and various iterations- total score will be taken and compared to PROMIS standards)
Change of erectile and sexual functions | Baseline- one year
  Testosterone Levels- measured in ng/dL (normal range 265-923 ng/dL)
Change of erectile and sexual functions | Baseline- one year
  FSH Levels- measured in mIU/mL (normal range 1.5-12.4 mIU/mL)
Change of erectile and sexual functions | Baseline- one year
  LH Levels- measured in IU/L (normal range 1.8-8.6 IU/L)
Change of erectile and sexual functions | Baseline- one year
  Prolactin Levels- measured in ng/mL (normal range <20 ng/mL)
Change of erectile and sexual functions | Baseline- one year
  Promise Bank V20 Erectile Function (11 total questions, ranging from almost never/never to almost always/always and various iterations-total score will be taken and compared to PROMIS standards)
Change of erectile and sexual functions | Baseline- one year
  Promis Scale V20 Interest In Sexual Activity (2 total questions ranging from not at all to very and never to always- total score will be taken and compared to PROMIS standards)
Change of erectile and sexual functions | Baseline- one year
  Promis 29 Profile V20 (29 total questions, ranging from not at all to very much and never to always- total score will be taken and compared to PROMIS standards)

CONTACTS AND LOCATIONS:
Overall Officials: Leshana St. Jean, PhD, Study Director — Vanderbilt University Medical Center
Locations (2):
- Nigeria (2):
  - Aminu Kano Teaching Hospital, Kano
  - Murtala Mohammed Specialist Hospital, Kano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piel FB, Hay SI, Gupta S, Weatherall DJ, Williams TN. Global burden of sickle cell anaemia in children under five, 2010-2050: modelling based on demographics, excess mortality, and interventions. PLoS Med. 2013;10(7):e1001484. doi: 10.1371/journal.pmed.1001484. Epub 2013 Jul 16. PMID 23874164
- [Background] Anele UA, Morrison BF, Burnett AL. Molecular pathophysiology of priapism: emerging targets. Curr Drug Targets. 2015;16(5):474-83. doi: 10.2174/1389450115666141111111842. PMID 25392014
- [Background] Huang AW, Muneyyirci-Delale O. Reproductive endocrine issues in men with sickle cell anemia. Andrology. 2017 Jul;5(4):679-690. doi: 10.1111/andr.12370. Epub 2017 Jun 29. PMID 28662541
- [Background] Adeyoju AB, Olujohungbe AB, Morris J, Yardumian A, Bareford D, Akenova A, Akinyanju O, Cinkotai K, O'Reilly PH. Priapism in sickle-cell disease; incidence, risk factors and complications - an international multicentre study. BJU Int. 2002 Dec;90(9):898-902. doi: 10.1046/j.1464-410x.2002.03022.x. PMID 12460353
- [Background] Emond AM, Holman R, Hayes RJ, Serjeant GR. Priapism and impotence in homozygous sickle cell disease. Arch Intern Med. 1980 Nov;140(11):1434-7. PMID 6159833
- [Background] Serjeant G, Hambleton I. Priapism in Homozygous Sickle Cell Disease: A 40-year Study of the Natural History. West Indian Med J. 2015 Jun;64(3):175-80. doi: 10.7727/wimj.2014.119. Epub 2015 Apr 27. PMID 26426165
- [Background] Virag R, Bachir D, Lee K, Galacteros F. Preventive treatment of priapism in sickle cell disease with oral and self-administered intracavernous injection of etilefrine. Urology. 1996 May;47(5):777-81; discussion 781. doi: 10.1016/s0090-4295(96)00027-1. PMID 8650886
- [Background] Okpala I, Westerdale N, Jegede T, Cheung B. Etilefrine for the prevention of priapism in adult sickle cell disease. Br J Haematol. 2002 Sep;118(3):918-21. doi: 10.1046/j.1365-2141.2002.03691.x. PMID 12181066
- [Background] Olujohungbe AB, Adeyoju A, Yardumian A, Akinyanju O, Morris J, Westerdale N, Akenova Y, Kehinde MO, Anie K, Howard J, Brooks A, Davis VA, Khoriatry AI. A prospective diary study of stuttering priapism in adolescents and young men with sickle cell anemia: report of an international randomized control trial--the priapism in sickle cell study. J Androl. 2011 Jul-Aug;32(4):375-82. doi: 10.2164/jandrol.110.010934. Epub 2010 Dec 2. PMID 21127308
- [Background] Rachid-Filho D, Cavalcanti AG, Favorito LA, Costa WS, Sampaio FJ. Treatment of recurrent priapism in sickle cell anemia with finasteride: a new approach. Urology. 2009 Nov;74(5):1054-7. doi: 10.1016/j.urology.2009.04.071. Epub 2009 Jul 17. PMID 19616292
- [Background] Abern MR, Levine LA. Ketoconazole and prednisone to prevent recurrent ischemic priapism. J Urol. 2009 Oct;182(4):1401-6. doi: 10.1016/j.juro.2009.06.040. Epub 2009 Aug 15. PMID 19683289
- [Background] DeCastro BJ, Costabile RA, McMann LP, Peterson AC. Oral ketoconazole for prevention of postoperative penile erection: a placebo controlled, randomized, double-blind trial. J Urol. 2008 May;179(5):1930-2. doi: 10.1016/j.juro.2008.01.039. Epub 2008 Mar 18. PMID 18353393
- [Background] Saad ST, Lajolo C, Gilli S, Marques Junior JF, Lima CS, Costa FF, Arruda VR. Follow-up of sickle cell disease patients with priapism treated by hydroxyurea. Am J Hematol. 2004 Sep;77(1):45-9. doi: 10.1002/ajh.20142. PMID 15307105
- [Background] Burnett AL, Bivalacqua TJ, Champion HC, Musicki B. Feasibility of the use of phosphodiesterase type 5 inhibitors in a pharmacologic prevention program for recurrent priapism. J Sex Med. 2006 Nov;3(6):1077-1084. doi: 10.1111/j.1743-6109.2006.00333.x. PMID 17100941
- [Derived] Idris IM, Yusuf AA, Ismail II, Borodo AM, Hikima MS, Kana SA, Aliyu T, Musangedu K, Jibrilla AU, Aji SA, Kuliya-Gwarzo A, Mohammad K, Galadanci JA, Alkassim R, Suwaid MA, Hussaini N, Rodeghier M, Burnett AL, DeBaun MR. A controlled trial for preventing priapism in sickle cell anemia: hydroxyurea plus placebo vs hydroxyurea plus tadalafil. Blood. 2025 Jun 26;145(26):3101-3112. doi: 10.1182/blood.2024027898. PMID 40073378

DOCUMENTS (1):
  • Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT05142254/ICF_000.pdf